CLINICAL TRIAL: NCT03390010
Title: Intrauterine Misoprostol With Active Management of Labour Versus Active Management of Labour for Prevebtion of Postpartum Hemorage in Cesarean Section ,Randomized Controlled Trial
Brief Title: Misoprostol Versus Active Management of Labour in CS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aljazeera Hospital (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Active management of labour
Record Dates: First submitted 2017-12-28; First posted 2018-01-04 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Cesarean Section
MeSH Terms: interventions — Misoprostol; Oxytocin; Methylergonovine; Carboprost; Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extra medication group (Active Comparator): -Procedure : Giving misoprostol plus syntocinon during CS
  this group in which prevention of uterine atony is made by intrauterine misoprostol plus the usual syntocinon and using extra uterotonic drugs when needed ; methergine , carboprost
  Interventions: Drug: Misoprostol + syntocinon and using extra uterotonic drugs when needed ; methergine
- Active management of labour group (Active Comparator): * Procedure: Giving syntocinon during cesarean section
  * this group in which prevention of uterine atony is made by the usual active management of labour syntocinon and using extra uterotonic drugs when needed ; methergine , carboprost
  Interventions: Drug: Syntocinon and using extra uterotonic drugs when needed ; methergine carboprost

INTERVENTIONS:
Drug: Misoprostol + syntocinon and using extra uterotonic drugs when needed ; methergine — medical prophylaxis against postpartum atony and postpartum hemorage by giving misoprostol plus syntocinon and using extra uterotonic drugs when needed ; methergine, carboprost
  Other Names: DrugsMisoprostol plus syntocinon and using extra uterotonic drugs when needed ; methergine , carboprost
  Arms: Extra medication group
Drug: Syntocinon and using extra uterotonic drugs when needed ; methergine carboprost — medical prophylaxis against postpartum atony and postpartum hemorage by giving syntocinon and using extra uterotonic drugs when needed ; methergine, carboprost
  Other Names: drugs ( syntocinon and using extra uterotonic drugs when needed ; methergine, carboprost
  Arms: Active management of labour group

SUMMARY:
Several treatment strategies are emplemented to prevent post delivery hemorage and decreasing maternal morbidity and mortality .

DETAILED DESCRIPTION:
Many approved drugs are used in prophylaxis against postpartum hemorage from these medications are the (syntocinon combined with methergine ) that are known as active management of labour drugs .

Moreover there is misotac , that also guards against postpartum hemorage .

All these medications act in a different way to cause uterine contraction post delivery to prevent uterine atony .

-Here we are comparing the additive value of misotac intrauterine to syntocinon and methergine in comparison to the usually used syntocinon plus methergine .

ELIGIBILITY:
Inclusion Criteria:

* • All patients included in this research were aged 18-42 years, pregnant 37 weeks till 42 weeks

  * no medical disorders with pregnancy e.g DM, HTN. All patients were subjected to full history taking, examination.

Exclusion Criteria:

* Exclusion Criteria:

  * The following patients were excluded , GA before 37 weeks or after 42 weeks , medical disorders with pregnancy eg. DM with pregnancy, HTN with pregnancy

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant females
Enrollment: 300 (Actual)
Dates: Start 2017-12-28 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-03-06 (Actual)

PRIMARY OUTCOMES:
The number of participants who passed cesarean section without postpartum hemorage | within 2 days post CS

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, M.s.c, Study Chair — Algazeerah hospital -Location (Giza -Egypt ); yossra Lasheen, M.D, Principal Investigator — kasraliny hospital- Aljazeerah hospital
Locations (1):
- Algazeerah, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No